CLINICAL TRIAL: NCT00333541
Title: Internet Access and Use in Women at High Risk for Unintended Pregnancy: A Randomized Clinical Trial
Brief Title: Evaluation of Internet Access and Use in Adolescent Women Initiating Contraception
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Health Services Research
Other Study IDs: R01HD045480-03 (NIH)
Record Dates: First submitted 2006-06-02; First posted 2006-06-05 (Estimated); Last update posted 2015-03-05 (Estimated); Status verified 2015-03

CONDITIONS: Contraceptive Behavior; Internet Use
Keywords: Contraceptive behavior; Internet Use; Adolescent pregnancy; Unintended pregnancy
MeSH Terms: conditions — Contraception Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment (Experimental): follow-up via e-mail link to survey
  Interventions: Behavioral: Using internet/E-mail for follow-up
- Control (No Intervention): standard follow-up by phone and in-person interview

INTERVENTIONS:
Behavioral: Using internet/E-mail for follow-up — follow-up via email link to survey
  Arms: Treatment

SUMMARY:
This purpose of this study is determine whether the use of internet technology to communicate with adolescents about contraception is feasible and to determine whether it is more effective than traditional methods. Study subjects will complete baseline and follow-up surveys at 3, 6, and 12 months about their contraceptive practice and sexual behaviors.

Subjects with internet access will be randomized to either completing surveys remotely over the internet through email or to follow-up in clinic on laptop computers.

Our hypothesis is that women who have access to the internet as well as use the internet regularly are more likely to complete follow-up surveys. This will then in turn allow us to get a better understanding of contraceptive practices amongst high risk teens.

DETAILED DESCRIPTION:
Despite the wide range of contraceptive technologies currently available the rate of unintended pregnancies in the U.S. remains high. In particular, adolescents, unmarried, low income, and minority women are amongst the highest risk populations for unintended pregnancy . Improving contraceptive use is critical for addressing this problem. Many programs have been developed and implemented to reduce sexual risk-taking behavior, one of the precursors to unintended pregnancies. Unfortunately, most of them have met with mixed results. Gaining insight into contraceptive practice and sexual behavior in this population is the first step towards improving contraceptive use. Many other disciplines have successfully used the internet for purposes of research (ie. asthma management, smoking cessation,etc), but this use of the internet has not been explored with adolescent women.

The study we are proposing is a randomized control trial to evaluate the use of internet technology in communicating with adolescent women about contraceptive practice. This study is a sub-study within an ongoing 12-month, longitudinal observational study of a cohort of "high-risk" women and their contraceptive practices and sexual behavior. Our hypothesis is that women who have access to the internet are more likely to complete follow-up surveys while enrolled in this longitudinal study, thus enabling us to obtain a greater understanding about contraceptive practice within this population via the internet. Furthermore, if internet proves to be a more effective means of communicating with adolescents because of the potential convenience and privacy of the method we may increase our impact on contraceptive use by embracing internet technology in the future.

Participants with internet access within the larger study will be identified and entered into a sub-study and randomized to either in clinic follow-up surveys or remote access completion of surveys via email over the internet. All participants will undergo the same screening, consent, and entry criteria for the study.

ELIGIBILITY:
Inclusion Criteria:

* Women age 15-24
* Sexually active
* Single
* Initiating contraception: either OCP's, the patch, the ring, or depoprovera
* English speaking
* Have an active email account
* Use email use ≥1 per wk

Exclusion Criteria:

* Lack of email account
* Email use < 1 per wk

Ages: 15 Years to 24 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 100 (Actual)
Dates: Start 2006-06; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Primary outcome: total # of subjects who complete all 3 follow-up surveys at 3, 6, and 12 months in each arm of the study | 1 year

SECONDARY OUTCOMES:
Secondary outcome: evaluate the feasibility of using internet technology in this population by looking at how many subjects actually has access to the internet and report regular use in the entire cohort | 1 year
and evaluate subject satisfaction with each method | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Tina Raine, MD, MPH, Principal Investigator — University of California, San Francisco; Sadia Haider, MD, MPH, Principal Investigator — University of California, San Francisco

REFERENCES:
- [Derived] Haider S, Dodge LE, Brown BA, Hacker MR, Raine TR. Evaluation of e-mail contact to conduct follow-up among adolescent women participating in a longitudinal cohort study of contraceptive use. Contraception. 2013 Jul;88(1):18-23. doi: 10.1016/j.contraception.2012.11.016. Epub 2013 Jan 3. PMID 23290427